CLINICAL TRIAL: NCT06765070
Title: Efficacy and Usability of the EXPLORER Exoskeleton in Children With Neurodevelopmental Disorders in Their Natural Environment
Brief Title: Efficacy and Usability of the EXPLORER Exoskeleton in Children With Neurodevelopmental Disorders in Natural Environments
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: MarsiBionics (Industry)
Collaborators: Hospital Infantil Universitario Niño Jesús, Madrid, Spain (Other); Hospital General Universitario Gregorio Marañon (Other); Hospital Universitario La Paz (Other); Hospital Universitario 12 de Octubre (Other); Universidad Rey Juan Carlos (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EXP-I-EF
Record Dates: First submitted 2024-12-20; First posted 2025-01-09 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Neuromuscular Disorders; Neurodevelopmental Disorders
Keywords: Neurodevelopmental disorders; Neuromuscular disorders; cerebral palsy; acquired brain injury; spinal muscular atrophy; robotics; gait; rehabilitation; spinal cord injury
MeSH Terms: conditions — Neuromuscular Diseases; Neurodevelopmental Disorders; Cerebral Palsy; Brain Injuries; Muscular Atrophy, Spinal; Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- EXPLORER (Experimental): Two-week period with the robotics gait device for use in the natural settings deemed appropriate by the family.
  Interventions: Device: EXPLORER

INTERVENTIONS:
Device: EXPLORER — Two-week period with the robotics gait device for use in the natural settings deemed appropriate by the family.

SUMMARY:
Neurodevelopmental disorders often lead to abnormal development of the Central Nervous System (CNS), frequently causing motor dysfunctions such as an inability to stand and walk. EXPLORER is a robotic gait exoskeleton designed to rehabilitate children with motor disabilities in home and outdoor environments.

The aim of this study is to evaluate the efficacy and usability of EXPLORER in children with motor disability within their natural settings, including home and community environments.

DETAILED DESCRIPTION:
Neurodevelopmental disorders often lead to abnormal development of the Central Nervous System (CNS), frequently causing motor dysfunctions such as an inability to stand and walk. Robotic devices are a useful tool in the rehabilitation of these children, but most of them are designed to be used in the clinical setting. EXPLORER is a robotic device designed to assist gait in children with motor disability in their homes and the community. The aim of this study is to evaluate the efficacy and usability of EXPLORER in children with motor disability within their natural settings, including home and community environments.

An initial session will be conducted in the participant's natural environment, during which the researchers will instruct the primary caregivers on the use of the device. Subsequently, the device will be left for a two-month period for use in the natural settings deemed appropriate by the family.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of any pathology or condition causing neurodevelopmental disorders.
* Ability to continuously use the device for two weeks, at least 3 times per week, without causing excessive fatigue that would prevent the participant from carrying out their usual activities.
* Availability and commitment from the family to use the device at least 3 times per week during the planned period, in different environments and with various objectives.
* Medical authorization for standing, gait training and weight bearing.
* Informed consent signed by legal guardians.
* Maximum user weight of 60 kg.
* Hip width (between greater trochanters) ≤37 cm.
* Length of the thigh (distance from the greater trochanter to the lateral condyle of the tibia) from 21cm to 36cm.
* Tibia leg length (distance from the lateral condyle of the tibia to the lateral malleolus) from 20cm to 35cm.
* Shoe size ≤40 (EU)

Exclusion Criteria:

* Medical contraindications for standing or walking.
* Non-reducible contractures or heterotropic ossifications above the degrees allowed by the device or out of the trajectory imposed by the device
* Spasticity equal to 4 on the Modified Ashworth Scale at the time of use of the device.
* More than 20º of hip and/or knee non-reducible contractures at the time of using the exoskeleton.
* Necessity to walk with more than 5º of hip abduction.
* Impossibility to reach 5º of ankle dorsiflexion with ir without orthoses.
* Lower length dysmetria that cannot be mitigated with a wedge under the foot.
* Skin lesion on parts of the lower extremities that are in contact with the device.
* History of fracture without trauma.
* Presence of other conditions causing exercise intolerance (such as uncontrolled hypertension, coronary artery disease, arrhythmia, congestive heart failure, severe pulmonary disease).
* Conductual disorders that may interfere with the use of the device or their participation in the study, like impulsiveness.
* Allergy to any of the EXPLORER materials: cotton, nylon, polyester, PPS, PEEK or ABS.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Serious Adverse Events | through study completion, along 2 weeks
  occurrence of any serious adverse event to the participant or the caregiver
Falls prevalence | through study completion, along 2 weeks
  Number of falling events occurred from the participant or caregiver
Skin integrity | through study completion, along 2 weeks
  Occurrence of any injury of the skin in the areas of contact and produced by the use of the device
Pain (Visual Analogic Scale) | through study completion, along 2 weeks
  pain measured by the Visual Analogic Scale (VAS) by the participant and the caregiver, scored from 0 to 10, being 0 "no pain" and 10 "unbearable pain"
Donning and doffing time | through study completion, along 2 weeks
  Time to don and doff the device to each participant
Device usage time | through study completion, along 2 weeks
  Time using the device
Number of steps | through study completion, along 2 weeks
  number of steps with the device
Usage modes | through study completion, along 2 weeks
  two different usage modes (active and automatic).
Speed | through study completion, along 2 weeks
  speed achieved with the device (steps per minute)
Device accessibility | through study completion, along 2 weeks
  Environments where the device has been used and level of accessibility in each environment measured with a 5 points Likert scale (0 not accessible - 5 very accessible)
Range of motion | Before starting the intervention (S1) and after completing the two weeks of use
  Passive Degree to which a joint can move (hip, knee, and ankle joints in both legs). From 0º to 180º.
Participation | Before starting the intervention (S1) and after completing the two weeks of use
  Measured with the Child and Adolescent Scale of Participation. 20 ordinal scaled items across 4 subsections.
  Maximum total score is 80 (20 items x 4) and the minimum total score is 20 (20 items x 1)

SECONDARY OUTCOMES:
QUEST | at the end of the intervention
  Using the Quebec User Evaluation of Satisfaction with Assistive Technology (QUEST 2.0) questionnaire administered to the participants' caregivers at the end of the intervention. The QUEST 2.0 scale has 12 items. Each item is rated on a 5-point Likert scale

CONTACTS AND LOCATIONS:
Locations (6):
- Spain (6):
  - Universidad Rey Juan Carlos, Alcorcón, Madrid
  - Hospital Universitario Gregorio Marañón, Madrid, Madrid
  - Hospital Infantil Universitario Niño Jesús - Servicio de Rehabilitación, Madrid, Madrid
  - Hospital Infantil Universitario Niño Jesús-Servicio de Neuro Ortopedia, Madrid, Madrid
  - Hospital Universitario 12 Octubre, Madrid, Madrid
  - Hospital Universitario La Paz, Madrid, Madrid